CLINICAL TRIAL: NCT01034735
Title: Phase I, Open Label, Randomised Three-way Cross Over, Single-centre Trial to Assess the Bioequivalence for Two Concentrations of the New r-hGH Liquid Multidose Formulation Versus the r-hGH Freeze-dried Multidose Formulation Administered in Healthy Volunteers
Brief Title: r-hGH Liquid Multidose Versus Freeze-dried Multidose Bioequivalence Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 28798
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Growth Failure; Growth Hormone Deficiency
Keywords: Saizen®; bioequivalence; recombinant human; Growth Hormone; treatment of growth failure in children; growth hormone deficiency in adults
MeSH Terms: conditions — Failure to Thrive; Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental)
  Interventions: Biological: r-hGH liquid (Saizen)
- Arm B (Experimental)
  Interventions: Biological: r-hGH liquid (Saizen)
- Arm C (Experimental)
  Interventions: Biological: r-hGH freeze-dried

INTERVENTIONS:
Biological: r-hGH liquid (Saizen) — Treatment Arm A: r-hGH liquid multidose formulation 5.83 mg/mL, needle injection (0.686 mL)
  Arms: Arm A
Biological: r-hGH liquid (Saizen) — Treatment Arm B: r-hGH liquid multidose formulation 8.0 mg/mL, needle injection (0.5 mL)
  Arms: Arm B
Biological: r-hGH freeze-dried — Treatment Arm C: r-hGH 8 mg (8.8 mg/1.51 ml) freeze-dried formulation ( reconstituted in metacresol 0.3% w/v) needle injection (0.686 mL)
  Arms: Arm C

SUMMARY:
The primary objective of the trial was to assess the bioequivalence for two concentrations (5.83 mg/mL and 8 mg/mL) of the new r-hGH liquid multidose formulation using the r hGH freeze-dried multidose formulation (Saizen® 8 mg, 8.8 mg/1.51 mL) as reference.

Each volunteer received three r hGH treatments, with each treatment being administered as a single subcutaneous dose of 4 mg r-hGH in a randomized sequence with at least one week of wash-out period between successive treatments.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

1. Male and female aged 18 to 45 years, inclusive; who are able to read, to write and to fully understand German language
2. Had given written Informed Consent
3. Had a body weight greater than 55 kg and a body mass index (BMI) of >20 and < or = 30 kg/m2 (BMI = weight (kg)/height (m)2)
4. Had vital signs in the following normal range:

   Ear body temperature: 35.0 - 38.0°C

   Blood pressure (BP) - after at least 3 minutes of rest, measured in the supine position:

   systolic blood pressure: 90 - 145 mmHg diastolic blood pressure : 50 - 95 mmHg Pulse rate (PR): after at least 3 minutes of rest, measured in the supine position: 40 90 bpm
5. Smoked less than 10 cigarettes per day, consented to smoke less than 5 cigarettes per day during the trial period and were able to refrain from smoking during the confinement period
6. Were able to communicate well with the Investigator and willing to comply with the requirements of the entire trial
7. Were willing to undergo pituitary down-regulation by intravenous infusion with somatostatin for 25 hours

   If female:
8. Had a negative serum pregnancy test within three weeks prior to trial start and a negative urine pregnancy test at the day before dosing
9. Were pre-menopausal and using an adequate method of non-hormonal contraception (2 barrier methods, or one barrier method with spermicide, or non-hormonal intrauterine device), sexual abstinence or females with vasectomised partners during the entire trial

Exclusion Criteria:

Main exclusion criteria:

1. Any surgical or medical condition, including findings in the medical history or in the pre trial assessments, that in the opinion of the Investigator, constituted a risk or a contraindication for the participation of the subject in the trial or that could have interfered with the trial objectives, conduct or evaluation
2. Had any clinically significant abnormal laboratory test results in the pre-trial safety laboratory tests or any clinically abnormal findings on the 12 leads resting electrocardiogram (ECG) that in the opinion of the Investigator may have increased the safety risk to the subject
3. Had positive results for drugs of abuse or alcohol test
4. Had positive results from serology examination for Hepatitis B surface antigen (HBsAg) (not due to vaccination), Hepatitis B core antibody (HBcAb) (if positive, was to be verified by test for anti-Hbc-IgM), Hepatitis C Virus (anti-HCV) and Human Immunodeficiency Virus (anti-HIV 1 and 2) at screening
5. History or presence of hypertension or other significant cardiovascular abnormalities
6. History or presence of cholelithiasis
7. Significant history or clinical evidence of auto-immune, gastrointestinal, haematological, hematopoietic, hepatic, neurological, pancreatic or renal disease
8. History or presence of diabetes
9. History or presence of tumors of the pituitary gland or hypothalamus
10. Definite or suspected personal history or family history of adverse drug reaction or hypersensitivity to drugs with a similar chemical structure to somatropin or somatostatin or its excipients, use of any chronic medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoints were the pharmacokinetic (PK) parameters of r-hGH: the area under the serum concentration-time curve from time zero to last detectable serum concentration (AUC0 t) and the maximum observed serum concentration (Cmax). | 24 hours post r hGH dose

SECONDARY OUTCOMES:
Secondary endpoints included further PK parameters. | 15 +/-3 days post last r hGH dose
Safety and tolerability were evaluated by adverse events (AEs), medical history, physical examination, vital signs, local tolerability, visual analog scale (VAS), ECG recordings, glycemia measurements and laboratory tests. | 15 +/-3 days post last r hGH dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lissy, MD, Principal Investigator — AAIPharma Deutschland GmbH & Co. KG
Locations (1):
- AAI Pharma Deutschland GmbH & Co. KG, Neu-Ulm, Germany

REFERENCES:
- [Derived] Liedert B, Forssmann U, Wolna P, Golob M, Kovar A. Comparison of the pharmacokinetics, safety and tolerability of two concentrations of a new liquid recombinant human growth hormone formulation versus the freeze-dried formulation. BMC Clin Pharmacol. 2010 Oct 20;10:14. doi: 10.1186/1472-6904-10-14. PMID 20961422